CLINICAL TRIAL: NCT00713843
Title: Effectiveness of Manual Therapy and Physical Therapy in Patients With Subacute and Chronic Non-specific Neck Pain. A Randomized Controlled Trial.
Brief Title: Effectiveness of Manual Therapy in Patients With Neck Pain.
Acronym: NECKproject
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Rob Oostendorp, emeritus professor Allied Heath Sciences, Radboud University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL21128.091
Record Dates: First submitted 2008-06-30; First posted 2008-07-14 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Neck Pain
Keywords: Neck Pain; Manuel Therapy Utrecht; Physiotherapy
MeSH Terms: conditions — Neck Pain | interventions — Exercise Therapy; Educational Status; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Manual Therapy Utrecht (Experimental): Manual Therapy Utrecht (MTU) During the first consultation the manual therapist enquires about the complaints of the patient. The manual therapist conducts a number of measurements according to protocol. During treatment preferred movements are executed by the manual therapist in the patient's joints. The treatment techniques used by the manual therapist are very gentle mobilizations, without high velocity thrust techniques and are in general painless. In Manual Therapy Utrecht (MTU) it is common to give advices and recommend exercises.
  A treatment session lasts between 30 and 60 minutes (repeated after one or two weeks). The maximum number of sessions is six.
  The manual therapist has a minimum of five years of working experience.
  Interventions: Other: Manual Therapy Utrecht
- 2 Physical Therapy - Exercise Therapy (Active Comparator): The physical therapist conducts a complaint related function examination. Treatment consist of active exercises, manual traction or stretching and massage. The aims of active exercises are improvement of strength, mobility and movement coordination. Specific mobilization techniques are not a part of physiotherapeutic treatment. Treatment sessions take place no more than twice a week with a maximum of nine sessions (approximately 30 minutes) with a minimum of twenty minutes on active exercise therapy combined with instruction.
  To prevent overlap with MTU (experimental arm), physical therapists are selected who are not (also) trained as manual therapists or have started this education.
  The physical therapist has at least five years of working experience.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Manual Therapy Utrecht — Manual Therapy (6 weeks).
  Other Names: joint mobilisation and manipulation; exercise therapy with instruction
  Arms: 1 Manual Therapy Utrecht
Other: Physical Therapy — Physical Therapy (six weeks).
  Other Names: exercise therapy with instruction; massagetherapy
  Arms: 2 Physical Therapy - Exercise Therapy

SUMMARY:
Background of the study: Manual Therapy applied to patients with non-specific neck pain has been investigated several times, both internationally and nationally. In the Netherlands different types of manual therapy treatment exist. Manual Therapy, as practiced under the Utrecht School, has not been subject of a randomized controlled trial. There is a need to evaluate the effectiveness of this type of manual therapy.

Objective of the study: This trial will investigate the effectiveness of Manual Therapy in the short and long-term up to 52 weeks in patient with (sub) acute (minimal two weeks) and chronic (maximum 52 weeks) since last episode of neck pain. Functional state, pain and global perceived effect are the outcome variables.

Study design: The study is a single blind randomized controlled trial.

Study population: Men and women aged 18 to 70 years old with neck pain for at least two weeks.

Intervention: The experimental group will be treated with manual therapy for a period of six weeks. The control group will be treated with physical therapy (usual care) also for a period of six weeks.

Primary study parameters / outcome of the study: Global Perceived Effect (GPE) and the Neck disability index (NDI-DV ) will be applied.

Secondary study parameters / outcome of the study: Visual Analogue Scale (VAS) for pain and SF36 (Quality of life). The Multidimensional Health Locus of Control(MHLC ), Credibility/Expectancy Questionnaire, Fear Avoidance Beliefs Questionnaire (FABQ-DLV) will also be measured.

DETAILED DESCRIPTION:
Detailed information about Manual Therapy according to the Utrecht School Manual Therapy (MTU)

MTU is based on assessing the patient's individual preference of functioning by documenting and interpreting their natural asymmetry in anatomical form, posture and movements. The normal asymmetry and variability of human form and movement function have been specified. Asymmetrical forms can be related to the asymmetrical movement function.

In addition to the general diagnostics, MTU is characterized by specific diagnostics. By means of this specific manual-therapeutic analysis the individual preference of functioning model of the patient is drawn up through analysis and interpretation of the individual asymmetry in form, posture and movement. Some explanations of the measurements and movements are: (preferred) hand folding; (preferred) arm folding; which eye is master eye; leg use in (preferred) kicking of a ball. The purpose here is to describe the optimal direction and position of movement axes for all joints according to this model.

When composing this model, firstly the individual characteristics (a number of preferred movements, a number of asymmetrical aspects of posture and form) are assessed. Documentation, notation and interpretation of these characteristics take place according to a protocol.

The objective of MTU is to optimize the positioning of movement axes in the joints. To achieve this, three-dimensional movements in the joints are executed repeatedly. To purpose fully position the movement axes the therapist should (repeatedly) perform passive joint movements with low velocity and high accuracy. In addition to examining the individual preference of movement, exploratory examination is carried out to recognize possible red flags and to determine the treatment indication.

Treatment is based on preferred movements found in the patient and the interpretation according to the protocol of these movements and not on the complaint of the patient. It is executed by applying passive articular movements in the spinal joints and the joints of the extremities. During this process physiological joint limitations are carefully observed; traction or high-velocity movements will not be applied, as may be the case in other forms of manual therapy.

The diagnostic examination of other forms of manual therapy focuses on joint function, stability, movement patterns, range of movement, and the severity of disorders. To diagnose the patients complaints, palpation of passive accessory and passive intervertebral movements are used. The results yield information as to tenderness (pain), restricted intersegmental motion (stiffness), and spasm (muscle tension).

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least two weeks of neck pain
* Last episode starts at a maximum of one year ago
* Age between 18 and 70 years
* Patient is willing to undergo the treatment
* Neck pain is mechanical and can be provocated by movements or postures of the neck
* Neck pain is the main problem to treat
* Neck pain may also give pain in the upper arm or cervicogenic headaches

Exclusion Criteria:

* Appearance of "red flags"
* Cervical surgery in the past
* Pregnancy
* Whiplash trauma
* Health conditions with may disturb the treatment or makes it impossible to undergo the treatment.
* Not enough understanding of the Dutch questionnaires
* Undergoing treatments like physical therapy, manual therapy, osteopathy, chiropraxis, acupuncture, other types of exercise therapy during the last three months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-09; Primary Completion 2013-05 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Global Perceived Effect (GPE), Neck disability index (NDI-DV ) | 0-3-7-13-26-52 weeks

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) or Numeric Rating Scale (NRS)for pain and SF36 (Quality of life). Multidimensional Health Locus of Control (MHLC), credibility/ expectancy, Fear Avoidance Beliefs Questionaire (FABQ-DLV) | 0-3-7-13-26-52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rob Oostendorp, Prof. dr., Study Chair — UMC St Radboud, IQ healthcare, Nijmegen
Locations (1):
- NECKproject.nl, Dordrecht, South Holland, Netherlands

REFERENCES:
- [Derived] Groeneweg R, Haanstra T, Bolman CAW, Oostendorp RAB, van Tulder MW, Ostelo RWJG. Treatment success in neck pain: The added predictive value of psychosocial variables in addition to clinical variables. Scand J Pain. 2017 Jan;14:44-52. doi: 10.1016/j.sjpain.2016.10.003. Epub 2016 Nov 2. PMID 28850429
- [Derived] Groeneweg R, van Assen L, Kropman H, Leopold H, Mulder J, Smits-Engelsman BCM, Ostelo RWJG, Oostendorp RAB, van Tulder MW. Manual therapy compared with physical therapy in patients with non-specific neck pain: a randomized controlled trial. Chiropr Man Therap. 2017 Apr 28;25:12. doi: 10.1186/s12998-017-0141-3. eCollection 2017. PMID 28465824
- [Derived] van Dongen JM, Groeneweg R, Rubinstein SM, Bosmans JE, Oostendorp RA, Ostelo RW, van Tulder MW. Cost-effectiveness of manual therapy versus physiotherapy in patients with sub-acute and chronic neck pain: a randomised controlled trial. Eur Spine J. 2016 Jul;25(7):2087-96. doi: 10.1007/s00586-016-4526-0. Epub 2016 Mar 21. PMID 27001136
- [Derived] Groeneweg R, Kropman H, Leopold H, van Assen L, Mulder J, van Tulder MW, Oostendorp RA. The effectiveness and cost-evaluation of manual therapy and physical therapy in patients with sub-acute and chronic non specific neck pain. Rationale and design of a Randomized Controlled Trial (RCT). BMC Musculoskelet Disord. 2010 Jan 24;11:14. doi: 10.1186/1471-2474-11-14. PMID 20096136